CLINICAL TRIAL: NCT07307040
Title: Construction of a Precision and Individualized Management Model for Diabetes With Integrated Traditional Chinese and Western Medicine
Brief Title: Precision Diabetes Management: Integrated East-West Approach
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xinhua Xiao, Chief physician, Peking Union Medical College Hospital
Other Study IDs: CXZH2024059
Record Dates: First submitted 2025-12-01; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Early-Onset Type 2 Diabetes
Keywords: Integrated Traditional Chinese and Western Medicine; Precision Management; Personalized Management; Early-Onset Type 2 Diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Integrated Traditional Chinese and Western Medicine Management
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
This project will leverage a large-scale cohort of early-onset type 2 diabetes patients to conduct innovative prospective clinical research. By integrating traditional Chinese medicine diagnostic information, clinical data, laboratory results, continuous glucose monitoring, genetic information, multi-omics data, and multi-modal monitoring data, and utilizing advanced data analysis methods such as deep learning, the project aims to establish a comprehensive monitoring, precise classification, and personalized diagnosis and treatment model-a holistic management approach integrating traditional Chinese and Western medicine for early-onset type 2 diabetes. This initiative is expected to enhance the management of early-onset type 2 diabetes, improve treatment outcomes and quality of life for affected patients, pioneer an innovative path for personalized integrated traditional Chinese and Western medicine management in this population, and promote the application of precision medicine in diabetes prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* The age at diabetes diagnosis is ≥18 years but <40 years.

Exclusion Criteria:

* The clinical diagnosis was type 1 diabetes, and at the time of enrollment, antibody levels or insulin/C-peptide results still supported the original diagnosis.

There were clear secondary factors contributing to hyperglycemia, such as Cushing's syndrome or pheochromocytoma.

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: The age at type 2 diabetes diagnosis is ≥18 years but <40 years.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Traditional Chinese Medicine Syndrome Score | Through study completion, an average of 3 months
HbA1c | Through study completion, an average of 3 months

SECONDARY OUTCOMES:
Triglycerides | Through study completion, an average of 3 months
High-Density Lipoprotein Cholesterol | Through study completion, an average of 3 months
Total Cholesterol | Through study completion, an average of 3 months
Fasting Blood Glucose | Through study completion, an average of 3 months
Low-Density Lipoprotein Cholesterol | Through study completion, an average of 3 months